CLINICAL TRIAL: NCT02915796
Title: Autologous CD133(+) Cells as an Adjuvant to Below the Knee Percutaneous Transluminal Angioplasty: A Randomized Controlled Clinical Trial in Diabetic Patients With Below the Knee Critical Limb Ischemia
Brief Title: Autologous CD133(+) Cells as an Adjuvant to Below the Knee Percutaneous Transluminal Angioplasty
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Maoquan Li, Prof. Dr. Li, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-xjs-08
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Endothelial progenitor cell; Percutaneous transluminal angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Granulocyte Colony-Stimulating Factor; AC133 Antigen; Cell Count; Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- G-CSF + CD133(+) cells + PTA (Experimental): Intramuscular injection of G-CSF along with transarterial infusion of CD133 (+) cells combined with percutaneous transluminal angioplasty
  Interventions: Biological: G-CSF + CD133(+) cells; Procedure: percutaneous transluminal angioplasty (PTA)
- PTA + G-CSF (Active Comparator): Percutaneous transluminal angioplasty along with intramuscular injection of G-CSF
  Interventions: Biological: G-CSF; Procedure: percutaneous transluminal angioplasty (PTA)
- Only PTA (Placebo Comparator): Only Percutaneous transluminal angioplasty along with placebo infusion of sodium chloride injection
  Interventions: Procedure: percutaneous transluminal angioplasty (PTA); Biological: Placebo infusion

INTERVENTIONS:
Biological: G-CSF + CD133(+) cells — Patients in the G-CSF + CD133(+) cells + PTA group, received 150 unit of recombinant human G-CSF intramuscular injection to mobilize CD 133 cells from bone marrow to peripheral blood. After 72-120 hrs, 100 ml suspension of peripheral arterial blood were collected and send to Good Products Manufacturing (GPM) certified laboratory (Shanghai Chen Chuan Biological Material Co. Ltd.) within 24 hrs of obtaining sample to isolate CD 133(+) endothelial progenitor cells (EPC) using magnetic cell separator. Subjects in this group, after vascular PTA treatment, received transarterial infusion of 50 ml suspension of isolated autologous CD 133(+) cells over 30 min via catheter opened into popliteal artery. The infusion of CD 133 cells was repeated after 24 hours.
  Arms: G-CSF + CD133(+) cells + PTA
Biological: G-CSF — Subjects in this group, after vascular PTA treatment, received 150 unit of recombinant human G-CSF intramuscular injection to mobilize EPCs from bone marrow to peripheral blood. But the C133 (+) cells were not isolated from the peripheral blood to infuse transarterially as in G-CSF + CD133(+) + PTA.
  Arms: PTA + G-CSF
Procedure: percutaneous transluminal angioplasty (PTA) — Subjects in this group only underwent below the knee percutaneous transluminal angioplasty .
Biological: Placebo infusion — Neither G-CSF was injected nor CD133(+) cells. Instead, subjects received placebo infusion (50 ml of 0.9% sodium chloride injection ) over 30 min.
  Arms: Only PTA

SUMMARY:
The main aim of the present study was to evaluate the therapeutic potential and safety of transarterial infusion of granulocyte colony stimulating factor (G-CSF) mobilized cluster of differentiation (CD) 133(+) cells when combined with percutaneous transluminal angioplasty (PTA) in treatment of below the knee (BTK) peripheral arterial disease (PAD) in diabetic patients.

DETAILED DESCRIPTION:
CD133+ cell, a bone marrow derived subpopulation of adult hematopoietic progenitor cells, confers high proliferative, vasculogenic and regenerative capacity in vitro and in vivo. thereby suggesting that CD133+ cells may induce vasculogenesis, improve limb perfusion, prevent tissue loss and restore ambulatory function in patients with critical limb ischemia. Although several small, randomized trials have been conducted so far demonstrating safety of autologous cells of bone marrow origin for the treatment, the reported benefits were found to be variable. A meta-analysis of autologous bone marrow derived cell therapy for critical limb ischemia trials suggested that application of autologous stem cell transplantation in curing limb ischemic patients does not have obviously effectiveness in the improvement of ankle brachial pressure (ABI) of the limb ischemic patients. But it can dramatically reduce the rate of amputation.

Therefore, in the present study, the investigators aim to evaluate the therapeutic potential and safety of transarterial infusion of g-csf-mobilized CD 133(+) cells when combined with PTA in treatment of below the knee PAD in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years , Gender: Both
2. Patients with below the knee limb ischemia with diabetes.
3. Rutherford class 2-6.
4. Target lesions with a diameter reduction of at least 50% and have an occlusion of longer than 4 cm on angiography.
5. Have no previous history of any stem cell therapy [infusion of CD133 endothelial progenitor cell (EPC)].

Written informed consent signed by the patients or representatives. -

Exclusion Criteria:

1. Previous bypass surgery or stent placement at the ipsilateral lower limb
2. History of intolerance to antiplatelet therapy, heparin, or contrast media.
3. Presence of any of the following conditions:

   1. severe liver disease (such as ascites, esophageal varices, liver transplantation);
   2. hemodynamic instability;
   3. Severely impaired renal function (serum creatinine level > 2.5 mg/dL).
   4. Receiving immunosuppressive therapy;
   5. History of decompensated heart failure (New York Heart Association class III or IV and level) or myocardial infarction, or heart bypass surgery;
   6. Bleeding diathesis;
   7. Active systemic bacterial infection;
   8. Acute thrombophlebitis or deep vein thrombosis of the target limb; 4) Pregnant or lactating women, or women of child bearing age unable or unwilling to use effective contraception during the study period; 5) Expected survival time of less than 24 months -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate | 12 months
  Occurrence of > 50% of restenosis in the treated vessel after 12 months as assessed by digital substraction angiography (DSA) (Efficacy endpoints).
Peak systolic velocity ratio | 12 months
  Peak systolic velocity ratio ≥ 2.4 by Doppler's ultrasonography for patients who did not undergo angiography after 12 months (Efficacy endpoints).
Severe adverse effects (SAEs) | 12 months
  Number of SAEs per subject across actual treatment cohorts (Safety Endpoint).

SECONDARY OUTCOMES:
ABI value | 6 and 12 months
  Improvement in ABI value by ≥ 0.1 after the procedure and lack of deterioration > 0.15 in relation to the maximal value recorded before the procedure.
Rutherford classification | 6 and 12 months
  improvement in Rutherford scale of at least one category after the procedure.
Transcutaneous oxygen pressures (TcPO2) | 6 and 12 months
  .Changes in TcPO2 was assessed at each follow up interval and compared to baseline.
Amputation-free survival (AFS) | 6 and 12 months
  Time to below the knee amputation of the ipsilateral leg.
Rest pain | 6 and 12 months
  Rest pain was measured using Wong-Baker FACES pain rating scale at baseline and each follow-up visit.
Six Minute Walk test | 6 and 12 months
  Walking distance, time to onset of leg cramping/pain were recorded.
Ulcer healing rate | 6 and 12 months
  Ulcer status was assessed at each follow up interval and compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Tong ji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma N, Ladilov Y, Moebius JM, Ong L, Piechaczek C, David A, Kaminski A, Choi YH, Li W, Egger D, Stamm C, Steinhoff G. Intramyocardial delivery of human CD133+ cells in a SCID mouse cryoinjury model: Bone marrow vs. cord blood-derived cells. Cardiovasc Res. 2006 Jul 1;71(1):158-69. doi: 10.1016/j.cardiores.2006.03.020. Epub 2006 Apr 3. PMID 16730684
- [Background] Gehling UM, Ergun S, Schumacher U, Wagener C, Pantel K, Otte M, Schuch G, Schafhausen P, Mende T, Kilic N, Kluge K, Schafer B, Hossfeld DK, Fiedler W. In vitro differentiation of endothelial cells from AC133-positive progenitor cells. Blood. 2000 May 15;95(10):3106-12. PMID 10807776
- [Background] Peichev M, Naiyer AJ, Pereira D, Zhu Z, Lane WJ, Williams M, Oz MC, Hicklin DJ, Witte L, Moore MA, Rafii S. Expression of VEGFR-2 and AC133 by circulating human CD34(+) cells identifies a population of functional endothelial precursors. Blood. 2000 Feb 1;95(3):952-8. PMID 10648408
- [Background] Friedrich EB, Walenta K, Scharlau J, Nickenig G, Werner N. CD34-/CD133+/VEGFR-2+ endothelial progenitor cell subpopulation with potent vasoregenerative capacities. Circ Res. 2006 Feb 17;98(3):e20-5. doi: 10.1161/01.RES.0000205765.28940.93. Epub 2006 Jan 26. PMID 16439688
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Esato K, Hamano K, Li TS, Furutani A, Seyama A, Takenaka H, Zempo N. Neovascularization induced by autologous bone marrow cell implantation in peripheral arterial disease. Cell Transplant. 2002;11(8):747-52. PMID 12588106
- [Background] Fadini GP, Avogaro A. Autologous transplantation of granulocyte colony-stimulating factor- mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2006 Feb;29(2):478-9; author reply 479-80. doi: 10.2337/diacare.29.02.06.dc05-1770. No abstract available. PMID 16482702
- [Background] Miyamoto K, Nishigami K, Nagaya N, Akutsu K, Chiku M, Kamei M, Soma T, Miyata S, Higashi M, Tanaka R, Nakatani T, Nonogi H, Takeshita S. Unblinded pilot study of autologous transplantation of bone marrow mononuclear cells in patients with thromboangiitis obliterans. Circulation. 2006 Dec 12;114(24):2679-84. doi: 10.1161/CIRCULATIONAHA.106.644203. Epub 2006 Dec 4. PMID 17145986
- [Background] Kawamoto A, Katayama M, Handa N, Kinoshita M, Takano H, Horii M, Sadamoto K, Yokoyama A, Yamanaka T, Onodera R, Kuroda A, Baba R, Kaneko Y, Tsukie T, Kurimoto Y, Okada Y, Kihara Y, Morioka S, Fukushima M, Asahara T. Intramuscular transplantation of G-CSF-mobilized CD34(+) cells in patients with critical limb ischemia: a phase I/IIa, multicenter, single-blinded, dose-escalation clinical trial. Stem Cells. 2009 Nov;27(11):2857-64. doi: 10.1002/stem.207. PMID 19711453
- [Background] Lu D, Chen B, Liang Z, Deng W, Jiang Y, Li S, Xu J, Wu Q, Zhang Z, Xie B, Chen S. Comparison of bone marrow mesenchymal stem cells with bone marrow-derived mononuclear cells for treatment of diabetic critical limb ischemia and foot ulcer: a double-blind, randomized, controlled trial. Diabetes Res Clin Pract. 2011 Apr;92(1):26-36. doi: 10.1016/j.diabres.2010.12.010. Epub 2011 Jan 8. PMID 21216483
- [Background] Losordo DW, Kibbe MR, Mendelsohn F, Marston W, Driver VR, Sharafuddin M, Teodorescu V, Wiechmann BN, Thompson C, Kraiss L, Carman T, Dohad S, Huang P, Junge CE, Story K, Weistroffer T, Thorne TM, Millay M, Runyon JP, Schainfeld R; Autologous CD34+ Cell Therapy for Critical Limb Ischemia Investigators. A randomized, controlled pilot study of autologous CD34+ cell therapy for critical limb ischemia. Circ Cardiovasc Interv. 2012 Dec;5(6):821-30. doi: 10.1161/CIRCINTERVENTIONS.112.968321. Epub 2012 Nov 27. PMID 23192920
- [Background] Sun X, Ying J, Wang Y, Li W, Wu Y, Yao B, Liu Y, Gao H, Zhang X. Meta-analysis on autologous stem cell transplantation in the treatment of limb ischemic. Int J Clin Exp Med. 2015 Jun 15;8(6):8740-8. eCollection 2015. PMID 26309525